CLINICAL TRIAL: NCT03455920
Title: Management of Sleep Apnea Patients by a Clinical Nurse (Supernurse)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Annie C Lajoie (Other)
Collaborators: Laval University (Other)
Responsible Party: Sponsor-Investigator, Annie C Lajoie, MD, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sleep Apnea Supernurse
Record Dates: First submitted 2017-12-20; First posted 2018-03-07 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Sleep Apnea Syndromes; Sleep Apnea; Multidisciplinary Communication; Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidisciplinary arm (Experimental): Patients randomized in this group will have their first sleep clinic evaluation with the clinical nurse. She will then discuss each case with the pulmonologist and validate the diagnostic and therapeutic avenue.
  Interventions: Other: Clinical nurse (supernurse) evaluation
- Pulmonologist arm (Active Comparator): Patients randomized in this group will have their first sleep clinic evaluation with the pulmonologist.
  Interventions: Other: Pulmonologist evaluation

INTERVENTIONS:
Other: Clinical nurse (supernurse) evaluation — The first evaluation of the patient refered to the sleep clinic will be performed by the clinical nurse then discussed with the pulmonologist in charge.
  Arms: Multidisciplinary arm
Other: Pulmonologist evaluation — The first evaluation of the patient refered to the sleep clinic will be performed only by the pulmonologist.
  Arms: Pulmonologist arm

SUMMARY:
Sleep apnea is a prevalent problem and references for the evaluation of this condition often exceeds the sleep clinic's capacity thus creating important delays in the patients' care.

The overall goal of this project is to assess the feasibility and the non-inferiority of integrating a clinical nurse, or supernurse, to the initial consultation team.

The hypothesis is that the integration of a clinical nurse to the sleep clinic's evaluation team is non inferior in terms of patients' outcomes such as improvement of symptoms and quality of life as well as adherence to treatment.

This study is supported by funding dedicated to teaching and research activities related to sleep-disordered breathing.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the ''Institut Universitaire de Cardiologie et Pneumologie de Québec'' 's sleep clinic who have undergone a cardiorespiratory polygraphy.
* Body mass index (BMI) between 27-35 kg/m2;
* Apnea-Hypopnea Index (ADI) equal or above 20 events per hour with less than 5 events per hour of central origin;
* Oxygen Desaturaton Index (ODI) equal or above 10 events per hour;
* Percentage of time spent below 90% of oxygen saturation equal or less than 10%

Exclusion criteria :

- Patients not meeting the above inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Improvement in symptoms | Assessed at three months
  Based on the Epworth Sleepiness scale (ranging from 0 to 24 points, higher values indicates increased sleepiness)
Improvement in symptoms | Assessed at six months
  Based on the Epworth Sleepiness scale (ranging from 0 to 24 points, higher values indicates increased sleepiness)

SECONDARY OUTCOMES:
Improvement in quality of life | Assessed at three months
  Based on the Quebec Sleep questionnaire
Improvement in quality of life | Assessed at six months
  Based on the Quebec Sleep Questionnaire
Positive pressure treatment adherence | Assessed at six months
  Number of hours used per night according to CPAP report
Mandibular advancement device treatment adherence | Assessed at six months
  According to the patient's usage report
Weight loss treatment adherence | Assessed at six months
  Changes from baseline weight (kg)
Positional therapy | Assessed at six months
  Proportion of time spent supine at baseline and at control cardio-respiratory recording

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Québec (CRIUCPQ), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antic NA, Buchan C, Esterman A, Hensley M, Naughton MT, Rowland S, Williamson B, Windler S, Eckermann S, McEvoy RD. A randomized controlled trial of nurse-led care for symptomatic moderate-severe obstructive sleep apnea. Am J Respir Crit Care Med. 2009 Mar 15;179(6):501-8. doi: 10.1164/rccm.200810-1558OC. Epub 2009 Jan 8. PMID 19136368
- [Background] Chai-Coetzer CL, Antic NA, Rowland LS, Reed RL, Esterman A, Catcheside PG, Eckermann S, Vowles N, Williams H, Dunn S, McEvoy RD. Primary care vs specialist sleep center management of obstructive sleep apnea and daytime sleepiness and quality of life: a randomized trial. JAMA. 2013 Mar 13;309(10):997-1004. doi: 10.1001/jama.2013.1823. PMID 23483174
- [Background] Robertson S, Maxwell C, McGarry GW, MacKenzie K. A nurse-led snoring clinic: how we do it. Clin Otolaryngol. 2009 Apr;34(2):158-61. doi: 10.1111/j.1749-4486.2009.01898.x. No abstract available. PMID 19413617
- [Background] Tomlinson M, John Gibson G. Obstructive sleep apnoea syndrome: a nurse-led domiciliary service. J Adv Nurs. 2006 Aug;55(3):391-7. doi: 10.1111/j.1365-2648.2006.03907.x. PMID 16866834
- [Background] Chai-Coetzer CL, Antic NA, Rowland LS, Catcheside PG, Esterman A, Reed RL, Williams H, Dunn S, McEvoy RD. A simplified model of screening questionnaire and home monitoring for obstructive sleep apnoea in primary care. Thorax. 2011 Mar;66(3):213-9. doi: 10.1136/thx.2010.152801. Epub 2011 Jan 20. PMID 21252389
- [Derived] Lajoie AC, Prive A, Roy-Halle A, Page D, Simard S, Series F. Diagnosis and management of sleep apnea by a clinical nurse: a noninferiority randomized clinical trial. J Clin Sleep Med. 2022 Jan 1;18(1):89-97. doi: 10.5664/jcsm.9502. PMID 34170235

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT03455920/Prot_SAP_000.pdf